CLINICAL TRIAL: NCT00667823
Title: Long-term Single-arm Open-label Extension Study of the SERAPHIN Study, to Assess the Safety and Tolerability of ACT 064992 in Patients With Symptomatic Pulmonary Arterial Hypertension
Brief Title: Clinical Study to Assess the Long-term Safety and Tolerability of ACT 064992 in Patients With Symptomatic Pulmonary Arterial Hypertension
Acronym: SERAPHIN OL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-055-303
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2022-02-10 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: SERAPHIN; Pulmonary Arterial Hypertension; ACT-064992
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — macitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ACT-064992 (Experimental): ACT-064992
  Interventions: Drug: Macitentan

INTERVENTIONS:
Drug: Macitentan — Tablet, oral administration, 10 mg dose once daily
  Other Names: ACT-064992

SUMMARY:
The main objective of the AC 055 303/SERAPHIN OL study, which will follow the AC 055 302/SERAPHIN study, will be to assess the long-term safety and tolerability of ACT 064992 in patients with symptomatic PAH.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to initiation of any study-mandated procedure.
* Patients with pulmonary arterial hypertension and having completed the event-driven study, AC 055 302/SERAPHIN, or Patients who have experienced a clinical worsening of PAH in AC 055 302/SERAPHIN and for whom a written approval to roll over into this study has been obtained from the Sponsor.
* Women of childbearing potential must have a negative pre-treatment serum pregnancy test and must use a reliable method of contraception during study treatment and for at least 28 days after study treatment termination.

Exclusion Criteria:

* Any major violation of protocol AC 055 302/SERAPHIN.
* Pregnancy or breast-feeding.
* AST and/or ALT > 3 times the upper limit of the normal range.
* Any known factor or disease that might interfere with treatment compliance, study conduct or interpretation of the results, such as drug or alcohol dependence or psychiatric disease.
* Known hypersensitivity to ACT 064992 or any of the excipients.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2008-10-17 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (158):
- United States (39):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Pulmonary Specialists, Phoenix, Arizona
  - University of California, San Diego, La Jolla, California
  - GLVA Healthcare Center, Los Angeles, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Liu Center for Pulmonary Hypertension, Torrance, California
  - University of Colorado CARDIAC AND VASCULAR CENTER, Aurora, Colorado
  - University of Florida - Division of Pulmonology, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - Emory University Hospital - McKelvey Center for Lung Transplantation & Pulmonary Vascular Disease, Atlanta, Georgia
  - Pulmonary & Critical Care of Atlanta, Atlanta, Georgia
  - Atlanta Institute for Medical Research, Decatur, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Iowa, Pulmonary Hypertension Program, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kentuckiana Pulmonary Associate, PLLC, Louisville, Kentucky
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Maryland School of Medicine; Division of Cardiology, Baltimore, Maryland
  - Pulmonary/Critical Care Division/Tufts New England Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Harper Univ. Hospital/ Wayne State University, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of NJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Columbia University Medical Center - Pediatric Cardiology, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Ohio Heart Health Center, Cincinnati, Ohio
  - Ohio State University, Div. of Pul. & Critical Care, Columbus, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Medical Center - St. Paul University, Dallas, Texas
  - Baylor College of Medicine and the Methodist Hospital,, Houston, Texas
  - University of Texas Houston Health Center, Houston, Texas
  - Intermountain Med Ctr- Pulm Dept Heart and Lung Ctr, Murray, Utah
  - Sentara Hospitals T/A Sentara Cardiovascular Research Intitute, Norfolk, Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Argentina (8):
  - Sanatorio Otamendi y Miroli S.A., Buenos Aires, Ciudad Autonoma
  - Hospital Britanico, Buenos Aires, Ciudad Autonoma
  - Sanatorio MITRE, Buenos Aires
  - Fundacion Favaloro, Buenos Aires
  - Instituto Cardiologia Corrientes, Corrientes
  - Htal Italiano Cordoba, Córdoba
  - Htla privado de Cordoba, Córdoba
  - Hospital Italiano - Garibaldi de Rosario, Santa Fe
- Australia (3):
  - St. Vincent's Hospital, Darlinghurst
  - The Alfred Hospital, Melbourne
  - Royal Brisbane Hospital, Sunshine Coast
- Medical University of Vienna/ Department of Internal Medicine II, Division of Cardiology, Vienna, Austria
- Belarus (3):
  - Republican reserach - Pratical Centre of Cardiology, Minsk
  - Minsk Regional Clinical Hospital, Minsk
  - Vitebsk Regional Clinical Hospital, Vitebsk
- University Hospital Gasthuisberg, Leuven, Belgium
- Mhat Nat Card Hosp - Pediatric Clinic, Sofia, BG, Bulgaria
- Canada (4):
  - Peter Lougheed Centre, Calgary, Alberta
  - London Health Sciences Centre, London, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - L'Hopital Laval, Sainte-Foy, Quebec
- Chile (3):
  - Hospital del Torax, Santiago
  - Pontificia Universidad Catolica de Chile, Santiago
  - Hospital San Juan de Dios, Santiago
- China (8):
  - Beijing Anzhen Hospital of the Capital University of Medical Sciences, Cardiology Department, Beijing
  - Peking Union Medical College Hospital, Rheumatology Department, Beijing
  - Guangdong General Hospital, Cardiology Department, Guangzhou
  - Jiangsu Province Hospital - Pneumology Department, Nanjing
  - Renji Hospital, Rheumatology Department, Shanghai
  - Zhongshan Hospital Fudan University, Cardiology Department, Shanghai
  - Renji Hospital, Cardiology Department, Shanghai
  - Shanghai Pulmonary Hospital Department of Pulmonary Circulation, Shanghai
- Colombia (2):
  - Fundacion Cardiovascular de Colombia, Floridablanca, Santander Department
  - Fundacion Clinica Shaio, Bogotá
- Clinical Hospital Center, Rijeka, Croatia
- Helsinki University Central Hospital, Helsinki, Finland
- France (3):
  - Hosp Bicetre - Dept Pulmo & Resp Intensive Care, Le Kremlin-Bicêtre
  - Hopital Arnaud de Villeneuve Service des Maladies Respiratoires, Montpellier
  - Hopital Haut-Leveque-Maison du Haut-Leveque, Pessac
- Germany (13):
  - Unfallkrankenhaus Berlin, Klinik für Innere Medizin, Berlin
  - Universität zu Köln, Medizinische Klinik III, Abteilung Kardiologie, Cologne
  - Medizinische Klinik und Poliklinik I Universitätsklinikum Carl Gustav Carus, Dresden
  - Universitätsklinikum Essen, Klinik für Kardiologie , Zentrum für Innere Medizin, Essen
  - Universitätsklinikums Gießen und Marburg GmbH / Medizinische Klinik und Poliklinik II, Innere Med. / Pneumologie, Giessen
  - Universität Greifswald / Klinik für Innere Medizin B,, Greifswald
  - Universitätsklinikum Hamburg-Eppendorf / Onkologie, Hämatologie und Knochenmarktransplantation mit Sektion Pneumologie, Hamburg
  - Medizinische Hochschule Hannover / Klinik für Pneumologie, Hanover
  - Thoraxklinik am Universitätsklinikum Heidelberg, Heidelberg
  - Universitätskliniken des Saarlandes / Medizinische Klinik und Poliklinik, Innere Medizin V, Homburg/Saar
  - Universtätsklinik Leipzig, Leipzig
  - Medizinische Klinik und Poliklinik I der Ludwig-Maximilians-Universität München / Klinikum Großhadern, Schwerpunkt Pneumologie, Munich
  - Universitatsklinikum Regensburg/Innere Medizin II, Regensburg
- Prince of Wales Hospital/ Division of Rheumatology, Department of Medicine & Therapeutics, Hong Kong, Hong Kong
- Hungary (4):
  - Gottsegen György Országos Kardiológiai Intézet (Hungarian Institute of Cardiology), Budapest
  - "Semmelweis Egyetem, Pulmonológiai Klinika", Budapest
  - University of Pecs, Medical School/Heart Institute and 1st Department of Internal Medicine, Pécs
  - University of Szeged Albert Szent-Gyorgyi Medical & Pharmaceutical Center, Szeged
- India (6):
  - Life Care Institute of Medical Science & Research, Ahmedabad, Ahmedabad
  - Care Hospital, Hyderabad
  - Seth GS Medical College & King Edward VII Memorial (KEM) Hospital / Department Of Cardiology, Mumbai
  - P D Hinduja National Hospital and Medical Research Centre/ Pulmunory Medicine, Mumbai
  - G B Pant Hospital & Maulana Azad Medical College, New Delhi
  - Deenanath Mangeshkar Hospital and Research Centre, Pune
- Israel (6):
  - Rambam Health Care Campus / Division of Medicine, Institute of Pulmonology, Haifa
  - Lady Davis Carmel Medical Center / Department of Cardiovascular Medicine, Pulmonary Division, Haifa
  - Rabin Medical Center - Belinson campus - Pulmonary Institute, Petach - Tikvah
  - Pulmonary Institute, Kaplan Medical Center, Rehovot
  - Sourasky Medical Center - Division of Pulmonary Medicine and Allergy, Tel Aviv
  - The pulmonary institute Sheba Medical centre, Tel Litwinsky
- Italy (2):
  - IRCCS Policlinico San Matteo Policlinico / Dipartimento di Cardiologia, Pavia
  - Policlinico Umberto I, Cardiologia, Roma
- Institut Jantung Negara (National Heart Institute), Kuala Lumpur, Malaysia
- Mexico (2):
  - Instituto Nacional de Cardiología (INC) Ignacio Chávez, Mexico City
  - Unidad de Investigación Clinica en Medicina, Monterrey
- Netherlands (2):
  - VU Medisch Centrum, Dept. Pulmonology 4A 48, Amsterdam
  - St. Antonius ziekenhuis, Nieuwegein
- Peru (3):
  - Hospital Alberto Sabogal Sologuren - EsSALUD, Callao
  - Clinica Medica Cayetano Heredia, Lima
  - Instituto de Enfermedades Respiratorias, Lima
- Poland (3):
  - Klinika Chorob Serca i Naczyn Instytut Kardiologii Collegium Medicum UJ, Krakow
  - Cardiology Otwock Priv, Otwock
  - III Katedra i Oddział Kliniczny Kardiologii Slaskiego Uniwersytetu Medycznego, Zabrze
- Romania (2):
  - Institutul de boli cardiovasculare / Clinica de Cardiologie, Bucharest
  - Institutul de Pneumologie "Marius Nasta" / I. Clinica de Pneumoftiziologie, Bucharest
- Russia (12):
  - Municipal Health Care Institution Kemerovo Cardiology Dispensary, Kemerovo
  - Federal State Institution "State Scientific Research Centre of Preventive Medicine" of Rosmedtechnology, Moscow
  - Federal State Institution "Scientific Research Institute of Pulmonology of Roszdrav", Moscow
  - State Health Care Institution of Moscow "City Clinical Hospital #1 named after N. I. Pirogov", Moscow
  - Federal State Institution "Russian Cardiology Scientific and Production Complex of Rosmedtechnology", Moscow
  - State Educational Institution "St Petersburg Medical Academy of Postgraduate Education" of Federal Agency of Public Health and Social Development, Saint Petersburg
  - State Educational Institution of High Professional Education "St Petersburg State Medical, Saint Petersburg
  - Federal State Institution "Federal Center of Heart, Blood and Endocrinology named after V.A. Almazov" of Rosmedtechnology, Saint Petersburg
  - State Institution "Scientific Research Institute of Cardiology" of Tomsk Scientific Center of RAMS, Siberian branch, Tomsk
  - Tomsk Regional Clinical Hospital / Pulmonology Unit, Tomsk
  - Municipal Health Care Institution "Clinical Hospital of Emergency Care named after N.V. Soloviov", Yaroslavl
  - Sverdlovsk Regional Clinical Hospital # 1/ Cardiology Department (2nd Therapy Department), Yekaterinburg
- Serbia (3):
  - University Children's Hospital (UNIVERZITETSKA DECJA KLINKIKA), Belgrade
  - University Clinical Center of Serbia/ Institute for Lung Diseases and Tuberculosis, Belgrade
  - Zemun Clinical Hospital (Klinicko-bolnicki centar Zemun) / Department of Cardiology, Belgrade
- Singapore (2):
  - National University Hospital/ The Heart Institute, Singapore
  - National Heart Centre (Nhc) Singapore, Singapore
- Slovakia (2):
  - National Institute of Cardiovascular Diseases (Slovenska zdravotnicka univerzita) / Faculty of Medical Specialty Studies (Fakulta zdravotnickych speci, Bratislava
  - Slovak Medical University (Slovenská zdravotnícka univerzita) / Faculty of Medical Speciality Studies (Fakulta zdravotníckych špecializačných štúdií), Bratislava
- South Africa (4):
  - Tread Research, Cape Town
  - Chris Hani Baragwanath Hospital, Department of Cardiology, Johannesburg
  - Netcare Milpark Hospital,Center for Chest Disease, Johannesburg
  - Block 4, Vergelegen Medi-Clinic, Somerset West
- Sweden (2):
  - University Hospital of Lund, Dept. of Cardiology, Lund
  - Uppsala University Hospital, Cardiology, Uppsala
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital/ Thoracic Surgical Division, Surgical Department, Taipei
- Thailand (4):
  - Ramathibodi Hospital, Mahidol University, Cardiology Unit, Department of Medicine,, Bangkok
  - Siriraj Hospital, Mahidol University, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Division of Rheumatology, Chiang Mai
  - Srinagarind Hospital/Division of Rheumatology, Department of Medicine, Faculty of Medicine, Khon Kaen University, Khon Kaen
- Ukraine (3):
  - Dnipropetrovsk State Medical Academy / Regional Diagnostic Center, Department of electrophysiologic researches and anaesthesiologic aid, Dnipro
  - Danylo Galytskyi Lviv State Medical University, Lviv
  - Odessa State Medical University, Military-medical Clinical Center of the South region, Odesa
- Royal Free Hospital, London, United Kingdom

REFERENCES:
- [Derived] Souza R, Delcroix M, Galie N, Jansa P, Mehta S, Pulido T, Rubin L, Sastry BKS, Simonneau G, Sitbon O, Torbicki A, Boyanova N, Chamitava L, Stein C, Channick RN. Long-Term Safety, Tolerability and Survival in Patients with Pulmonary Arterial Hypertension Treated with Macitentan: Results from the SERAPHIN Open-Label Extension. Adv Ther. 2022 Sep;39(9):4374-4390. doi: 10.1007/s12325-022-02199-x. Epub 2022 Jul 12. PMID 35819570
- [Derived] Krause A, Zisowsky J, Dingemanse J. Modeling of pharmacokinetics, efficacy, and hemodynamic effects of macitentan in patients with pulmonary arterial hypertension. Pulm Pharmacol Ther. 2018 Apr;49:140-146. doi: 10.1016/j.pupt.2018.02.005. Epub 2018 Feb 28. PMID 29501590

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant flow reported below is up to study closure.
Groups:
- Macitentan 10 mg: Participants with symptomatic pulmonary arterial hypertension (PAH) who completed or have experienced a morbidity/clinical worsening of PAH in the study AC-055-302 (NCT00660179) and opted to continue this open label extension (OLE) study received macitentan oral tablet, 10 milligrams (mg) once daily from Day 1 up to end of study (up to 12 years) which depends on following a). transition to commercially available macitentan in the participant's country b). the sponsor decided to stop the OL study, and c). the participant's or investigators or sponsors decision to discontinue study treatment.
Period: Overall Study
Arm/Group | Macitentan 10 mg
Started | 550
Completed | 334
Not Completed | 216
Not completed — Lost to Follow-up | 5
Not completed — Adverse Event | 7
Not completed — Death | 182
Not completed — Withdrawal by Subject | 12
Not completed — Other | 8
Not completed — Missing (completion page missing) | 2

BASELINE CHARACTERISTICS:
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 550
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (15.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 440
  Male | 110
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 165
  Other | 13
  White | 372
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 32
  AUSTRALIA | 6
  AUSTRIA | 4
  BELARUS | 21
  BELGIUM | 2
  BULGARIA | 4
  CANADA | 12
  CHILE | 24
  CHINA | 74
  COLOMBIA | 7
  FRANCE | 8
  GERMANY | 27
  HONG KONG | 3
  HUNGARY | 4
  INDIA | 30
  ISRAEL | 10
  ITALY | 3
  MALAYSIA | 6
  MEXICO | 33
  NETHERLANDS | 1
  PERU | 4
  POLAND | 19
  ROMANIA | 12
  RUSSIAN FEDERATION | 54
  SERBIA | 13
  SINGAPORE | 12
  SLOVAKIA | 4
  SOUTH AFRICA | 17
  SWEDEN | 6
  TAIWAN | 14
  THAILAND | 19
  UKRAINE | 12
  UNITED KINGDOM | 4
  UNITED STATES | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) up to 28 Days After Study Treatment Discontinuation
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAE are defined as AEs with onset during the treatment period or that are a consequence of a pre-existing condition that has worsened since baseline.
Time Frame: Up to 28 days after study treatment discontinuation (Up to 12 years)
Population: The safety analysis set (SAF) included all participants who received at least 1 dose of macitentan 10 milligrams (mg).
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 550
Participants | 527

2. Primary Outcome: Number of Participants With Death up to 28 Days After Study Treatment Discontinuation
Description: Number of participants with deaths up to 28 days after study treatment discontinuation were reported.
Time Frame: Up to 28 days after study treatment discontinuation (Up to 12 years)
Population: The SAF included all participants who received at least 1 dose of macitentan 10 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 550
Participants | 175

3. Primary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (TESAEs) up to 28 Days After Study Treatment Discontinuation
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAE are defined as AEs with onset during the treatment period or that are a consequence of a pre-existing condition that has worsened since baseline. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically significant, or requires intervention to prevent at least one of the outcomes listed above.
Time Frame: Up to 28 days after study treatment discontinuation (Up to 12 years)
Population: The SAF included all participants who received at least 1 dose of macitentan 10 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 550
Participants | 354

4. Primary Outcome: Number of Participants With AEs Leading to Permanent Discontinuation of Study Treatment
Description: Number of participants with AEs leading to permanent discontinuation of study treatment were reported. An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Up to 28 days after study treatment discontinuation (Up to12 years)
Population: The safety analysis set (SAF) included all participants who received at least 1 dose of macitentan 10 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 550
Participants | 62

5. Primary Outcome: Number of Participants With Treatment Emergent Abnormal Liver Tests up to 28 Days After Study Treatment Discontinuation
Description: Number of participants with treatment-emergent abnormal liver tests: Alanine aminotransferase (ALT) greater than (>) 3*upper limit of normal (ULN) or aspartate aminotransferase (AST) >3* ULN, ALT >5* ULN or AST >5*ULN, ALT >8*ULN or AST >8*ULN, total bilirubin (TBIL) >2*ULN, ALT >3*ULN or AST >3*ULN and TBIL >2*ULN at any time were reported.
Time Frame: Up to 28 days after study treatment discontinuation (Up to12 years)
Population: The SAF included all participants who received at least 1 dose of macitentan 10 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 550
Participants
  ALT or AST >3*ULN | 45
  ALT or AST >5*ULN | 20
  ALT or AST >8*ULN | 11
  TBIL >2*ULN | 75
  ALT or AST >3*ULN and (TBIL>2*ULN at any time) | 8

6. Primary Outcome: Number of Participants With Treatment Emergent Hemoglobin Abnormality up to 28 Days After Study Treatment Discontinuation
Description: Number of participants with treatment-emergent hemoglobin (HGB) abnormality up to 28 days after study treatment discontinuation were reported. Participants assessed for different categories of HGB were <=80 grams/Liter (g/L), <=100g/L, decrease from baseline >=20 g/L, and decrease from baseline >=50 g/L.
Time Frame: Up to 28 days after treatment discontinuation (Up to 12 years)
Population: The SAF included all participants who received at least 1 dose of macitentan 10 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 550
Participants
  HGB <= 80 gram/Liter (g/L) | 33
  HGB <= 100 g/L | 98
  HGB decrease from baseline >= 20 g/L | 188
  HGB decrease from baseline >= 50 g/L | 29

ADVERSE EVENTS:
Time Frame: Up to end of treatment plus 28 days for serious and other (non-serious) adverse events (Up to 11 years) and up to end of study for all-cause mortality (Up to 12 years)
Description: The safety analysis set (SAF) included all participants who received at least 1 dose of macitentan 10 milligrams (mg).
Arm/Group | Macitentan 10 mg
All-Cause Mortality (participants affected / at risk) | 182/550
Serious Adverse Events (participants affected / at risk) | 354/550
Other Adverse Events (participants affected / at risk) | 476/550
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan 10 mg (N=550)
Anaemia (Blood and lymphatic system disorders) | 27
Autoimmune Haemolytic Anaemia (Blood and lymphatic system disorders) | 1
Coagulopathy (Blood and lymphatic system disorders) | 1
Hypercoagulation (Blood and lymphatic system disorders) | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 3
Acute Coronary Syndrome (Cardiac disorders) | 1
Acute Myocardial Infarction (Cardiac disorders) | 2
Acute Right Ventricular Failure (Cardiac disorders) | 11
Angina Pectoris (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 3
Atrial Fibrillation (Cardiac disorders) | 7
Atrial Flutter (Cardiac disorders) | 8
Bradycardia (Cardiac disorders) | 1
Cardiac Arrest (Cardiac disorders) | 9
Cardiac Disorder (Cardiac disorders) | 1
Cardiac Failure (Cardiac disorders) | 7
Cardiac Failure Acute (Cardiac disorders) | 2
Cardiac Failure Chronic (Cardiac disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 6
Cardio-Respiratory Arrest (Cardiac disorders) | 4
Cardiogenic Shock (Cardiac disorders) | 9
Cardiopulmonary Failure (Cardiac disorders) | 2
Cardiorenal Syndrome (Cardiac disorders) | 1
Chronic Right Ventricular Failure (Cardiac disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 1
Cyanosis (Cardiac disorders) | 1
Left Ventricular Dysfunction (Cardiac disorders) | 1
Left Ventricular Failure (Cardiac disorders) | 2
Myocardial Infarction (Cardiac disorders) | 4
Myocardial Ischaemia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 3
Pericardial Effusion (Cardiac disorders) | 1
Right Ventricular Dysfunction (Cardiac disorders) | 1
Right Ventricular Failure (Cardiac disorders) | 72
Stress Cardiomyopathy (Cardiac disorders) | 1
Supraventricular Tachycardia (Cardiac disorders) | 2
Tachyarrhythmia (Cardiac disorders) | 1
Ventricular Fibrillation (Cardiac disorders) | 2
Ventricular Tachycardia (Cardiac disorders) | 1
Vertigo Positional (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Anal Fistula (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 3
Duodenal Perforation (Gastrointestinal disorders) | 1
Enterocolitis Haemorrhagic (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastritis Erosive (Gastrointestinal disorders) | 1
Gastroduodenitis (Gastrointestinal disorders) | 1
Gastrointestinal Disorder (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3
Gastrointestinal Necrosis (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Hiatus Hernia (Gastrointestinal disorders) | 1
Ileus Paralytic (Gastrointestinal disorders) | 1
Intestinal Pseudo-Obstruction (Gastrointestinal disorders) | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis Acute (Gastrointestinal disorders) | 2
Pancreatitis Relapsing (Gastrointestinal disorders) | 1
Peptic Ulcer (Gastrointestinal disorders) | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 2
Umbilical Hernia (Gastrointestinal disorders) | 3
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 2
Cardiac Death (General disorders) | 1
Chest Discomfort (General disorders) | 3
Chest Pain (General disorders) | 11
Death (General disorders) | 5
Drug Ineffective (General disorders) | 1
Fatigue (General disorders) | 2
General Physical Health Deterioration (General disorders) | 1
Influenza Like Illness (General disorders) | 1
Infusion Site Pain (General disorders) | 1
Multiple Organ Dysfunction Syndrome (General disorders) | 4
Oedema Peripheral (General disorders) | 2
Peripheral Swelling (General disorders) | 2
Pyrexia (General disorders) | 4
Sudden Cardiac Death (General disorders) | 3
Sudden Death (General disorders) | 11
Vascular Stent Thrombosis (General disorders) | 1
Bile Duct Stone (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis Acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 2
Hepatic Steatosis (Hepatobiliary disorders) | 1
Drug Hypersensitivity (Immune system disorders) | 1
Abscess Limb (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 3
Arthritis Bacterial (Infections and infestations) | 1
Atypical Pneumonia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 9
Bronchitis Viral (Infections and infestations) | 1
Candida Sepsis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 4
Device Related Infection (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 4
Gastroenteritis Bacterial (Infections and infestations) | 1
Gastroenteritis Norovirus (Infections and infestations) | 1
Gastroenteritis Salmonella (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Hiv Infection (Infections and infestations) | 2
Infected Skin Ulcer (Infections and infestations) | 2
Infective Exacerbation of Chronic Obstructive Airways Disease (Infections and infestations) | 1
Influenza (Infections and infestations) | 5
Joint Tuberculosis (Infections and infestations) | 1
Laryngitis Bacterial (Infections and infestations) | 1
Localised Infection (Infections and infestations) | 1
Lower Respiratory Tract Infection (Infections and infestations) | 8
Lung Infection (Infections and infestations) | 8
Meningitis (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumococcal Sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 40
Pneumonia Influenzal (Infections and infestations) | 1
Pneumonia Klebsiella (Infections and infestations) | 1
Pneumonia Streptococcal (Infections and infestations) | 1
Postoperative Wound Infection (Infections and infestations) | 1
Pulmonary Sepsis (Infections and infestations) | 2
Pulmonary Tuberculosis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Pyelonephritis Acute (Infections and infestations) | 2
Respiratory Tract Infection (Infections and infestations) | 3
Respiratory Tract Infection Viral (Infections and infestations) | 1
Salmonella Sepsis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 4
Septic Shock (Infections and infestations) | 6
Staphylococcal Bacteraemia (Infections and infestations) | 1
Subcutaneous Abscess (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 8
Urinary Tract Infection (Infections and infestations) | 3
Urosepsis (Infections and infestations) | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 1
Acetabulum Fracture (Injury, poisoning and procedural complications) | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 1
Brain Contusion (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 5
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1
Femur Fracture (Injury, poisoning and procedural complications) | 2
Foot Fracture (Injury, poisoning and procedural complications) | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 2
Perineal Injury (Injury, poisoning and procedural complications) | 1
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 2
Radius Fracture (Injury, poisoning and procedural complications) | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1
Subarachnoid Haemorrhage (Injury, poisoning and procedural complications) | 3
Subdural Haematoma (Injury, poisoning and procedural complications) | 2
Thermal Burn (Injury, poisoning and procedural complications) | 1
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 2
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 3
Traumatic Haematoma (Injury, poisoning and procedural complications) | 1
Traumatic Haemorrhage (Injury, poisoning and procedural complications) | 1
Ulna Fracture (Injury, poisoning and procedural complications) | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1
Anticoagulation Drug Level above Therapeutic (Investigations) | 1
Blood Bilirubin Increased (Investigations) | 1
Catheterisation Cardiac (Investigations) | 2
Computerised Tomogram Abnormal (Investigations) | 1
International Normalised Ratio Increased (Investigations) | 3
Investigation (Investigations) | 1
Liver Function Test Increased (Investigations) | 3
Oxygen Saturation Decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Electrolyte Imbalance (Metabolism and nutrition disorders) | 2
Fluid Overload (Metabolism and nutrition disorders) | 4
Fluid Retention (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 5
Metabolic Acidosis (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1
Mixed Connective Tissue Disease (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2
Polymyositis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 3
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 5
Systemic Scleroderma (Musculoskeletal and connective tissue disorders) | 2
Anogenital Warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cardiac Valve Fibroelastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastatic Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nasopharyngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectosigmoid Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Richter's Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous Cell Carcinoma of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous Cell Carcinoma of the Cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Amnesia (Nervous system disorders) | 1
Brain Oedema (Nervous system disorders) | 1
Cerebellar Infarction (Nervous system disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Hepatic Encephalopathy (Nervous system disorders) | 1
Ischaemic Stroke (Nervous system disorders) | 2
Loss of Consciousness (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 2
Radiculopathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 20
Abortion Missed (Pregnancy, puerperium and perinatal conditions) | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 2
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2
Device Dislocation (Product Issues) | 1
Device Malfunction (Product Issues) | 1
Anxiety (Psychiatric disorders) | 1
Anxiety Disorder (Psychiatric disorders) | 1
Completed Suicide (Psychiatric disorders) | 1
Confusional State (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Mental Status Changes (Psychiatric disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 8
Calculus Urinary (Renal and urinary disorders) | 1
Chronic Kidney Disease (Renal and urinary disorders) | 1
Cystitis Haemorrhagic (Renal and urinary disorders) | 1
Lupus Nephritis (Renal and urinary disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 1
Neurogenic Bladder (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Prerenal Failure (Renal and urinary disorders) | 1
Renal Colic (Renal and urinary disorders) | 3
Renal Failure (Renal and urinary disorders) | 2
Renal Impairment (Renal and urinary disorders) | 2
Ureterolithiasis (Renal and urinary disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Menometrorrhagia (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 2
Metrorrhagia (Reproductive system and breast disorders) | 1
Ovarian Cyst (Reproductive system and breast disorders) | 4
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 1
Ovarian Cyst Torsion (Reproductive system and breast disorders) | 1
Pelvic Haematoma (Reproductive system and breast disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Uterine Haemorrhage (Reproductive system and breast disorders) | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 1
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 123
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 10
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 6
Pulmonary Hypertensive Crisis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5
Respiratory Tract Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1
Aortic Surgery (Surgical and medical procedures) | 1
Bunion Operation (Surgical and medical procedures) | 1
Chemotherapy (Surgical and medical procedures) | 1
Cholecystectomy (Surgical and medical procedures) | 1
Gastric Polypectomy (Surgical and medical procedures) | 1
Hysterectomy (Surgical and medical procedures) | 1
Lung Transplant (Surgical and medical procedures) | 7
Oophorectomy (Surgical and medical procedures) | 1
Osteosynthesis (Surgical and medical procedures) | 1
Therapy Cessation (Surgical and medical procedures) | 1
Transfusion (Surgical and medical procedures) | 1
Accelerated Hypertension (Vascular disorders) | 1
Aneurysm Ruptured (Vascular disorders) | 1
Aortic Aneurysm (Vascular disorders) | 1
Aortic Aneurysm Rupture (Vascular disorders) | 1
Circulatory Collapse (Vascular disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 2
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 3
Hypovolaemic Shock (Vascular disorders) | 1
Venous Thrombosis Limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan 10 mg (N=550)
Anaemia (Blood and lymphatic system disorders) | 80
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 14
Leukopenia (Blood and lymphatic system disorders) | 22
Thrombocytopenia (Blood and lymphatic system disorders) | 36
Atrial Fibrillation (Cardiac disorders) | 24
Palpitations (Cardiac disorders) | 34
Right Ventricular Failure (Cardiac disorders) | 24
Tachycardia (Cardiac disorders) | 22
Hypothyroidism (Endocrine disorders) | 21
Abdominal Distension (Gastrointestinal disorders) | 14
Abdominal Pain (Gastrointestinal disorders) | 12
Abdominal Pain Upper (Gastrointestinal disorders) | 22
Constipation (Gastrointestinal disorders) | 20
Diarrhoea (Gastrointestinal disorders) | 59
Dyspepsia (Gastrointestinal disorders) | 13
Gastritis (Gastrointestinal disorders) | 11
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 21
Nausea (Gastrointestinal disorders) | 28
Vomiting (Gastrointestinal disorders) | 24
Chest Pain (General disorders) | 35
Fatigue (General disorders) | 19
Oedema Peripheral (General disorders) | 105
Pyrexia (General disorders) | 25
Hyperbilirubinaemia (Hepatobiliary disorders) | 26
Bronchitis (Infections and infestations) | 78
Cellulitis (Infections and infestations) | 11
Cystitis (Infections and infestations) | 11
Gastroenteritis (Infections and infestations) | 16
Influenza (Infections and infestations) | 17
Laryngitis (Infections and infestations) | 11
Lower Respiratory Tract Infection (Infections and infestations) | 12
Nasopharyngitis (Infections and infestations) | 105
Pharyngitis (Infections and infestations) | 28
Pneumonia (Infections and infestations) | 29
Respiratory Tract Infection (Infections and infestations) | 31
Respiratory Tract Infection Viral (Infections and infestations) | 23
Rhinitis (Infections and infestations) | 16
Sinusitis (Infections and infestations) | 18
Tooth Abscess (Infections and infestations) | 11
Upper Respiratory Tract Infection (Infections and infestations) | 121
Urinary Tract Infection (Infections and infestations) | 46
Ligament Sprain (Injury, poisoning and procedural complications) | 11
Alanine Aminotransferase Increased (Investigations) | 22
Aspartate Aminotransferase Increased (Investigations) | 20
Blood Bilirubin Increased (Investigations) | 16
Blood Creatinine Increased (Investigations) | 12
Haemoglobin Decreased (Investigations) | 13
Liver Function Test Increased (Investigations) | 15
Weight Decreased (Investigations) | 19
Decreased Appetite (Metabolism and nutrition disorders) | 18
Gout (Metabolism and nutrition disorders) | 16
Hyperglycaemia (Metabolism and nutrition disorders) | 11
Hyperkalaemia (Metabolism and nutrition disorders) | 16
Hyperuricaemia (Metabolism and nutrition disorders) | 15
Hypokalaemia (Metabolism and nutrition disorders) | 39
Arthralgia (Musculoskeletal and connective tissue disorders) | 33
Back Pain (Musculoskeletal and connective tissue disorders) | 33
Myalgia (Musculoskeletal and connective tissue disorders) | 15
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 12
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 21
Dizziness (Nervous system disorders) | 55
Headache (Nervous system disorders) | 63
Syncope (Nervous system disorders) | 40
Anxiety (Psychiatric disorders) | 13
Depression (Psychiatric disorders) | 12
Insomnia (Psychiatric disorders) | 36
Acute Kidney Injury (Renal and urinary disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 74
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 54
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 27
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 18
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 14
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 18
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 47
Rash (Skin and subcutaneous tissue disorders) | 16
Skin Ulcer (Skin and subcutaneous tissue disorders) | 13
Hypotension (Vascular disorders) | 20

LIMITATIONS AND CAVEATS:
The limitation of the open-label study design was the open label nature of the trial due to which the number of participants decreased over time to the extent that 10 percent (%) and 2.4% of participants (N=550) remained in the study at Years 7 and 9, respectively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT00667823/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/23/NCT00667823/SAP_001.pdf